CLINICAL TRIAL: NCT06809426
Title: Evaluating the Safety and Efficacy of 177Lu-LNC1011 Injection in a Single-Center, Single-Arm, Open Study in Patients with Prostate-Specific Membrane Antigen (PSMA)-Positive Metastatic Desmoplasia-Resistant Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS2023057
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: PSMA PET-Positive Castration-Resistant Prostate Cancer
Keywords: PSMA; mCRPC; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-LNC1011 (Experimental): Successfully screened subjects will be treated with 177Lu-LNC1011 Injection during the treatment period with 75 mCi (2.78 GBq) intravenously every 6 weeks for a total of no more than 6 doses. Subjects will be monitored for safety and anti-tumor efficacy after dosing during the treatment period.
  Interventions: Drug: 177Lu-LNC1011

INTERVENTIONS:
Drug: 177Lu-LNC1011 — 75 mCi (2.78 GBq) of 177Lu-LNC1011 Injection intravenously each time, injections every 6 weeks, not to exceed a total of 6 injections.

SUMMARY:
Evaluating the safety and antitumor efficacy of 177Lu-LNC1011

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, open IIT clinical study evaluating the safety and anti-tumor efficacy of 177Lu-LNC1011 Injection in patients with PSMA-positive metastatic desmoplasia-resistant prostate cancer (mCRPC). Thirteen patients are expected to be enrolled. Subjects will be required to sign an informed consent form prior to screening, and successful screened subjects will be treated with 177Lu-LNC1011 Injection as 75 mCi (2.78 GBq) intravenously every 6 weeks for a total of no more than 6 doses during the treatment period. Subjects will be monitored for safety and anti-tumor efficacy after dosing during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male.
2. histologically or cytologically defined prostate cancer, the patients have not been treated or have exhausted all treatment.
3. meet the Prostate Cancer Working Group 3 (PCWG3) diagnosis of metastatic desmoplasia-resistant prostate cancer (mCRPC), including: a) the presence of a desmoplasia level of serum testosterone (serum testosterone <50 ng/dL or 1.7 nmol/L); b) and the presence of one of the following: - serum PSA progression: PSA >1 ng/mL and 2 consecutive rises in PSA 1 week apart, 2 greater than 50% of the nadir; or a bone scan suggestive of ≥2 new bone lesions; or CT or MRI suggestive of progression of soft tissue lesions (RECIST 1.1).
4. a physical status score of ≤2 according to Eastern Cooperative Oncology Group (ECOG) criteria.
5. PSMA positivity confirmed by 68Ga -PSMA PET/CT.

Exclusion Criteria:

Patients who did not meet the requirements as assessed by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
To assess the difference in PSA changes before and after receiving 177Lu-LNC1011 treatment | 2-12 weeks
Objective remission rates in mCRPC patients as assess by RECIST V1.1 treated with 177Lu-LNC1011 | 2-12 weeks

SECONDARY OUTCOMES:
The radiation dose of 177Lu-LNC1011 in normal organs and tumors as assess by OLINDA/EXM | 1 day
The change of SUV (SUVmax, SUVmean) in 68Ga-PSMA PET/CT imaging before and after receiving 177Lu-LNC1011 treatment as assess by PMOD version 4.3 | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Affiated Hospital of Jiangnan University, Wuxi, Jiangsu, China

REFERENCES:
- [Derived] Hou L, Wang Y, Fu H, Chen L, Yu C, Chen X, Zhang J. PSMA-targeted radioligand therapy with [177Lu]Lu-LNC1011 for metastatic castration-resistant prostate cancer: a pilot study. Eur J Nucl Med Mol Imaging. 2025 Sep;52(11):4033-4043. doi: 10.1007/s00259-025-07245-8. Epub 2025 Apr 10. PMID 40208314